CLINICAL TRIAL: NCT04925141
Title: Efficacy and Safety of Dasatinib in the First-line Treatment of Newly Diagnosed Chronic-Phase Chronic Myeloid Leukemia (CML-CP)
Brief Title: A Study of Dasatinib as First-line Treatment for Newly Diagnosed Chronic-Phase Chronic Myeloid Leukemia (CML-CP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YNS-2015-V1.0
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib tablets (Experimental): Dasatinib tablets 100 mg orally once daily
  Interventions: Drug: Dasatinib Tablets

INTERVENTIONS:
Drug: Dasatinib Tablets — Tyrosine Kinase Inhibitor (TKI)

SUMMARY:
The purpose of this multicenter,open, prospective and single arm study is to evaluate the efficacy and safety of domestic dasatinib in the first-line treatment of newly diagnosed CML-CP.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and gender is not limited.
2. The chronic-phased CML subjects with Ph + were definitely diagnosed within 6 months before the first use of the study drug. The diagnostic criteria refer to the 2016 edition of Chinese CML diagnosis and treatment guidelines.
3. The Eastern Cooperative Oncology Group (ECOG) performance of 0-2.
4. The function of main organs such as liver and kidney is normal, which shows that serum bilirubin is less than or equal to 1.5 × ULN； Serum ALT and AST ≤ 2.5 × ULN； Serum Cr ≤ 1.5 × ULN； Serum amylase and lipase ≤ 1.5 × ULN; Blood potassium, magnesium, phosphorus and total calcium were more than or equal to the lower limit of normal value, or were corrected to normal range before administration.
5. The subjects voluntarily participate in and signed the informed consent form (ICF), and the process of signing the ICF meet the requirements of the "Practice for quality management of drug clinical trials".

Exclusion Criteria:

1. Subjects who have received any TKI treatment in the past.
2. Subjects who have received or are receiving anti CML chemotherapy drugs (except hydroxyurea).
3. Subjects who have received major surgery or no recovery from previous surgery within 4 weeks (including 4 weeks) before the first use of the study drug.
4. Subjects with mental illness, including epilepsy, dementia, severe depression, mania, etc.
5. Subjects with a history of significant congenital or acquired hemorrhagic disease unrelated to CML.
6. Disease history and comorbidities: a) uncontrolled severe disease or active infection that impairs the subject's ability to receive the treatment; b) Uncontrolled or major cardiovascular disease; c) Pulmonary hypertension; d) Subjects with pleural effusion or pericardial effusion of any grade are excluded when screening; when entering the study, subjects with remission of pleural / pericardial effusion of any grade previously diagnosed were allowed to participate in the study.
7. Subjects with gastrointestinal dysfunction or gastrointestinal diseases that may significantly affect the absorption of the test drug, such as ulcers, uncontrollable nausea, vomiting, diarrhea, malabsorption syndrome, after a small bowel resection, etc.
8. Cardiac dysfunction, including: a) complete left bundle branch block; b) Long QT syndrome, or known family history of long QT syndrome; c) Ventricular or atrial tachyarrhythmia of clinical significance; d) Clinically significant resting bradycardia (< 50 beats per minute); e) QTc>450msec； f) History of clinically confirmed myocardial infarction in the past 12 months; g) History of unstable angina in the past 12 months; h) Other clinicallysignificant heart diseases (e.g., congestive heart failure, etc.).
9. Combined with other primary malignant tumors (except basal cell carcinoma of skin).
10. Subjects who are receiving treatment with strong CYP3A4 inhibitors (e.g., erythromycin Ethylsuccinate, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, imipradil, etc.) and cannot discontinue or switch to other drugs before starting the study drug.
11. Subjects who are receiving strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampicin, rifabutin, rifapentine, phenobarbital, Hypericum perforatum, etc.) and the treatment cannot be stopped or replaced by other drugs before starting the study drug.
12. Subjectswho are receiving the treatment of drugs that may prolong QT interval, and the treatment can not be stopped or replaced by other drugs before starting to use the study drug.
13. Previous history of acute (within 1 year before inclusion) or chronic pancreatitis.
14. Known or suspected to be allergic to this kind of drug.
15. Female and male subjects of childbearing age who cannot use adequate methods of contraception , including pregnant or lactating women.
16. Subjects who are receiving the treatment of other test drugs or participated in the clinical trial of other drugs within one month.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve and maintain major molecular response (MMR) at 12 months | up to 12 months
  MMR is defined as BCR-ABL1IS ≤ 0.1%

SECONDARY OUTCOMES:
Proportion of subjects who achieve and maintain MMR at 3，6 and 18 months | up to 18 months
  MMR is defined as BCR-ABL1IS ≤ 0.1%
Time to MMR Overall | up to 24 months
  The time to MMR for all participants is defined as the time from first use of the study drug until measurement criteria are first met for MMR.
Cumulative MMR rates at 6, 12 and 24 months | up to 24 months
  MMR is defined as BCR-ABL1IS ≤ 0.1%
Proportion of subjects who achieve and maintain MR4.0 and MR4.5 at 6, 12 and 24 months | up to 24 months
  MR4.0 is defined as BCR-ABL1IS ≤ 0.01%, MR4.5 is defined as BCR-ABL1IS ≤ 0.0032%
Cumulative complete cytogenic response (CCyR) rates at 12 and 24 months | up to 24 months
  CCyR is defined as 0% Ph+ metaphases
Proportion of subjects who achieve and maintain complete hematological response (CHR) at 3 months | up to 3 months
  CHR was defined as peripheral blood WBC < 10x109 / L, PLT < 450x109 / L, no immature granulocytes, basophils < 0.05, no symptoms and signs of CML, spleen untouchable
Time to accelerated phase (AP ) / blast crisis (BC) | up to 24 months
  Time to AP / BC is defined as the time from the first use of the study drug to the date of CML related death or progression to AP or BC, whichever occurs first. For subjects without these events, the event was truncated at the date of the last evaluation (Hematology, extramedullary disease, or cytogenetic evaluation)
Progression-free Survival (PFS) | up to 24 months
  PFS is defined as the time from the first use of the study drug to the earliest occurrence of the following events: death from any cause (if death was the main cause of discontinuation) or progression to AP or BC.
Event free survival (EFS) | up to 24 months
  EFS is defined as the time from the first use of the study drug to the earliest occurrence of the following events during the study treatment: loss of CHR, loss of PCyCR, loss of CCyR, death from any cause during the treatment, and progression to AP or BC
ABL mutation rate after 6 months of treatment | up to 6 months
  The proportion of ABL mutations in subjects with BCR-ABL1IS > 1% or disease progression after 6 months of treatment
Incidence of adverse events (AEs) and serious adverse events (SAEs) to dasatinib | up to 24 months
  Evaluation of AEs, SAEs, and clinically relevant changes in laboratory tests according to laboratory reference ranges

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Affiliated Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Medical College , Zhejiang University, Hangzhou, Zhejiang